CLINICAL TRIAL: NCT01426672
Title: Monovision for Treatment of Diplopia
Brief Title: Monovision for the Treatment of Diplopia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mount Sinai Hospital, Canada (Other)
Responsible Party: Edward Margolin, MD, Mount Sinai Hospital
Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 08-0289-EMargolin
Record Dates: First submitted 2011-08-11; First posted 2011-08-31 (Estimated); Last update posted 2011-08-31 (Estimated); Status verified 2011-01

CONDITIONS: Strabismic Deviation
Keywords: Strabismic deviation less than 12 prism diopeters
MeSH Terms: interventions — Contact Lenses

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Monovision Correctoin (Experimental): Monovision correction
  Interventions: Other: Monovision Correction (with the help of glasses or contact lenses)

INTERVENTIONS:
Other: Monovision Correction (with the help of glasses or contact lenses)

SUMMARY:
PURPOSE:

The purpose of this study is to quantitatively assess the efficacy of monovision correction in the treatment of acquired small angle binocular diplopia in adult patients.

METHOD:

Twenty patients with symptomatic diplopia were enrolled in a prospective treatment trial. All had stable deviations of 10 prism diopters or less for over three months. Each received monovision spectacles and/ or contact lenses with distance correction in the dominant eye. Half received a +3.00 diopter (D) add and the others received +2.50 D. The validated and standardized Diplopia Questionnaire and Amblyopia and Strabismus Questionnaire (ASQE) were used to quantify the efficacy of monovision correction for diplopia by measuring the functional impact on vision-specific quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Strabismic Deviation less than 12 Prism Diopters

Exclusion Criteria:

* Inability to sign informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2009-01; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Patients satisfaction with monovision was measured by standardized diplopia questionnaire and results reported in statistical terms on multiple measures tested on the questionnaire. | 2 years
  To determine whether monovision correction was useful for the correction of small angle deviations in strabismic patients

CONTACTS AND LOCATIONS:
Locations (1):
- Edward Margolin, MD, Toronto, Ontario, Canada